CLINICAL TRIAL: NCT07229963
Title: Postprandial Cardiometabolic Effects of Interrupting Sedentary Behavior With Exercise of Varying Intensity in Healthy Overweight Adults
Brief Title: Exercise Intensity and Postprandial Effects of Breaking Sedentary Behavior in Overweight Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muhammed Mustafa Atakan, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SBA 25/679
Record Dates: First submitted 2025-09-24; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Risk Markers; Substrate Oxidation; Postprandial Metabolism; Exercise Physiology
Keywords: Exercise; Sedentary behavior; Cardiometabolic health; Postprandial metabolism; overweight
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary: Participants will remain seated for 7 h. (Experimental): The sedentary condition will take place in a seated position. During the seated condition, volunteers will be seated at a typical desk chair at an appropriate height with hip and knee angles of ~90° and feet flat on the floor. The seating area will include a standard desk chair, a work desk, and the volunteers' personal laptops. Volunteers will be instructed prior to the visit to avoid behaviors such as fidgeting, excessive leg movements, and crossing their legs to minimize potential extraneous effects.
  Interventions: Other: Sedentary Behaviour Intervention
- Breaking up sitting with aerobic exercise interruptions (Experimental): The protocol that will interrupt sitting with AEI will involve cycle exercises performed at 50% of VO2max for 2 minutes. The W and rpm levels corresponding to 50% of VO2max will be determined using the values recorded during the determination of VO2max.
  Interventions: Other: Aerobic Exercise Intervention
- Breaking up sitting with sprint exercise interruptions (Experimental): The protocol that will interrupt sitting with SEI will involve cycle exercises performed at the maximum revolutions per minute achievable within 10 seconds. Immediately before each SEI, volunteers will increase their pedal cadence to the maximum speed they can achieve, after which a pedal load will be applied to the bicycle ergometer and a sprint will be performed against the applied load for 10 seconds. During each sprint, the pedal load will be applied at 0.065 kilograms per kilogram of lean body mass. Since it has been shown to lead to greater peak power output in overweight and obese groups, lean body mass will be used as a reference when determining pedal load, rather than total body mass.
  Interventions: Other: Sprint Exercise Intervention

INTERVENTIONS:
Other: Aerobic Exercise Intervention — In the aerobic exercise condition, participants will perform 2 minutes of moderate-intensity continuous cycling.
  Arms: Breaking up sitting with aerobic exercise interruptions
Other: Sprint Exercise Intervention — In the sprint condition, participants will complete a 10-second all-out sprint, as determined during the preliminary test.
  Arms: Breaking up sitting with sprint exercise interruptions
Other: Sedentary Behaviour Intervention — Participants will remain seated for a total duration of 7 hours. During this period, they will be instructed to minimize excessive movement and will only be permitted to rise from the chair for voiding purposes.
  Arms: Sedentary: Participants will remain seated for 7 h.

SUMMARY:
The purpose of this study is twofold: (1) to determine whether breaking up prolonged sitting with aerobic or sprint cycling breaks reduces postprandial blood glucose, insulin, CRP, and blood pressure, which are established risk markers for cardiometabolic diseases; and (2) to assess substrate oxidation during this period in order to identify which exercise condition promotes the greatest increase in fat oxidation.

DETAILED DESCRIPTION:
Sedentary behavior (SED) refers to activities such as sitting, lying down, or reclining that require energy expenditure of ≤1.5 MET during the time spent awake. Prolonged and continuous sedentary behavior leads to adverse effects such as abnormal postprandial metabolic responses, insulin resistance, vascular dysfunction, high blood pressure, increased carbohydrate oxidation, and inflammation. Epidemiological data also show that SED increases the risk of mortality, cardiovascular disease, type 2 diabetes, and certain types of cancer. Experimental studies have shown that 2-5 minutes of low- or moderate-intensity aerobic exercise performed every 20-30 minutes during the postprandial period improves cardiometabolic health by reducing glucose, insulin, and blood pressure during the postprandial period. On the other hand, it is known that short-term sprint interval exercise (SIE) increases insulin sensitivity by rapidly depleting muscle glycogen, improves glucose control, lowers blood pressure, and increases fat oxidation. With these effects, SIE may be a time-efficient method for interrupting SED. Although the cardiometabolic benefits of SIE and aerobic exercise interruptions (AEI) are known, there is a lack of studies comparing the effects of interrupting SED with these two exercise types of different intensities in preventing postprandial cardiometabolic dysfunction. In this context, the aim of the study is to compare the postprandial cardiometabolic effects of interrupting sedentary behavior with AIE and sprint exercise interruptions (SEI) in overweight but otherwise healthy women and men aged 35-45. In this randomized crossover trial, volunteers will participate in three trials: 1) AEI, 2) SEI, and 3) SED. There will be a minimum 3-day washout period between trials. In the SEI and AEI trials, exercise interruptions will be implemented every 30 minutes during the 7-hour sitting period, whereas in the SED trial, participants will remain seated continuously for the entire duration. In all conditions, two meals (breakfast and lunch) will be served 3 hours apart, and the trials will begin, after the breakfast meal is consumed. Venous blood samples taken hourly during the experiment will be used to analyze insulin, glucose, and C-reactive protein (CRP) levels. In addition, blood pressure will be measured hourly, and fat oxidation will be assessed at the baseline, 2nd, 5th, and 7th hours. The effects of the conditions on glucose and insulin will be evaluated using linear mixed models. A Two-Way (Trial x Number of Repeats) Analysis of Variance for Repeated Measures will be used to detect differences between conditions.

ELIGIBILITY:
Inclusion Criteria

* Being physically inactive (not doing at least 150 minutes/week of structured exercise).
* Having a physical activity level of <5000 steps/day.
* Having a BMI between 25 and 29.9 kg/m2.
* Having a history of regular menstrual cycles for female participants.
* Having medical examination approval.

Exclusion Criteria

* Taking any acute or chronic medication or supplement that may affect metabolism.
* Having an acute or chronic illness that limits exercise (musculoskeletal problems, cardiovascular disorders, respiratory problems, etc.).
* Consuming tobacco products.
* Meeting 3 or more of the metabolic syndrome criteria (waist circumference of 102 cm or more in men, 88 cm or more in women, triglyceride level of 150 mg/dL or higher, HDL cholesterol level below 40 mg/dL in men and 50 mg/dL in women, blood pressure of 130/85 mmHg or higher, fasting blood glucose level of 100 mg/dL (5.6 mg/L) or higher).

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Insulin | 7 hour for each experimental condition
  Postprandial insulin. Net incremental area under the curve and total area under the curve for each 7 h condition will be calculated for insulin.

SECONDARY OUTCOMES:
Glucose | 7 hour for each experimental condition
  Postprandial glucose. Net incremental area under the curve and total area under the curve for each 7 hour condition will be calculated for glucose.
CRP | 7 hour
  Postprandial CRP. Net incremental area under the curve and total area under the curve for each 7 h condition will be calculated for CRP.
Substrate oxidation | 0, 2th, 5th, 7th hours
  Postprandial substrate oxidation. During each experimental visit, for 7 hours, volunteers' respiratory data will be collected using a direct calorimeter in a seated position for 10 minutes at 0, 2th, 5th, and 7th hours. The volunteers' resting fat and carbohydrate oxidations will be determined from the obtained data.
Blood pressure | 7 hour
  Postprandial arterial blood pressure will be measured hourly for 7 h using an automatic blood pressure monitor with a cuff of appropriate size. The systolic and diastolic BP values measured will be recorded, and the mean arterial pressure will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Nazan Koşar, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Sports Science Faculty, Hacettepe Beytepe Clinic, Ankara, Beytepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers due to privacy concerns and ethical restrictions outlined in the study's informed consent procedure.

REFERENCES:
- [Background] Compher C, Frankenfield D, Keim N, Roth-Yousey L; Evidence Analysis Working Group. Best practice methods to apply to measurement of resting metabolic rate in adults: a systematic review. J Am Diet Assoc. 2006 Jun;106(6):881-903. doi: 10.1016/j.jada.2006.02.009. PMID 16720129
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] DeMers D, Wachs D. Physiology, Mean Arterial Pressure. 2023 Apr 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538226/ PMID 30855814
- [Background] Stergiou GS, Palatini P, Parati G, O'Brien E, Januszewicz A, Lurbe E, Persu A, Mancia G, Kreutz R; European Society of Hypertension Council and the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement. J Hypertens. 2021 Jul 1;39(7):1293-1302. doi: 10.1097/HJH.0000000000002843. No abstract available. PMID 33710173
- [Background] Mattes RD, Campbell WW. Effects of food form and timing of ingestion on appetite and energy intake in lean young adults and in young adults with obesity. J Am Diet Assoc. 2009 Mar;109(3):430-7. doi: 10.1016/j.jada.2008.11.031. PMID 19248858
- [Background] Augustin LSA, Kendall CWC, Jenkins DJA, Willett WC, Astrup A, Barclay AW, Bjorck I, Brand-Miller JC, Brighenti F, Buyken AE, Ceriello A, La Vecchia C, Livesey G, Liu S, Riccardi G, Rizkalla SW, Sievenpiper JL, Trichopoulou A, Wolever TMS, Baer-Sinnott S, Poli A. Glycemic index, glycemic load and glycemic response: An International Scientific Consensus Summit from the International Carbohydrate Quality Consortium (ICQC). Nutr Metab Cardiovasc Dis. 2015 Sep;25(9):795-815. doi: 10.1016/j.numecd.2015.05.005. Epub 2015 May 16. PMID 26160327
- [Background] Diet, nutrition and the prevention of chronic diseases. World Health Organ Tech Rep Ser. 2003;916:i-viii, 1-149, backcover. PMID 12768890
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Carrillo-Arango HA, Atencio-Osorio MA, Lopez-Alban CA, Nava-Gonzalez EJ, Correa-Rodriguez M, Izquierdo M, Ramirez-Velez R. Metabolic responses to acute sprint interval exercise training performed after an oral 75-gram glucose load in individuals with overweight/obesity. Physiol Rep. 2023 Jan;11(2):e15555. doi: 10.14814/phy2.15555. PMID 36695728
- [Background] Ramirez-Velez R, Carrillo-Arango HA, Atencio-Osorio MA, Lopez-Alban CA, Calderon-Gonzalez JC, Morales-Alamo D, Izquierdo M, Correa-Rodriguez M. No sex differences in systemic metabolic responses to acute sprint interval training performed after an oral 75-g glucose load in adults with excess adiposity. Clin Nutr ESPEN. 2025 Feb;65:25-35. doi: 10.1016/j.clnesp.2024.11.005. Epub 2024 Nov 17. PMID 39551347
- [Background] Baker JS, Davies B. Brief high-intensity exercise and resistive force selection in overweight and obese subjects: body mass or body composition? Res Sports Med. 2006 Apr-Jun;14(2):97-106. doi: 10.1080/15438620600651298. PMID 16869135
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Midgley AW, McNaughton LR, Polman R, Marchant D. Criteria for determination of maximal oxygen uptake: a brief critique and recommendations for future research. Sports Med. 2007;37(12):1019-28. doi: 10.2165/00007256-200737120-00002. PMID 18027991
- [Background] Lanzi S, Codecasa F, Cornacchia M, Maestrini S, Salvadori A, Brunani A, Malatesta D. Fat oxidation, hormonal and plasma metabolite kinetics during a submaximal incremental test in lean and obese adults. PLoS One. 2014 Feb 11;9(2):e88707. doi: 10.1371/journal.pone.0088707. eCollection 2014. PMID 24523934
- [Background] Tudor-Locke C, Craig CL, Thyfault JP, Spence JC. A step-defined sedentary lifestyle index: <5000 steps/day. Appl Physiol Nutr Metab. 2013 Feb;38(2):100-14. doi: 10.1139/apnm-2012-0235. Epub 2012 Nov 8. PMID 23438219
- [Background] Schmidt MD, Cleland VJ, Shaw K, Dwyer T, Venn AJ. Cardiometabolic risk in younger and older adults across an index of ambulatory activity. Am J Prev Med. 2009 Oct;37(4):278-84. doi: 10.1016/j.amepre.2009.05.020. PMID 19765498
- [Background] Ekmekcioglu C, Touitou Y. Chronobiological aspects of food intake and metabolism and their relevance on energy balance and weight regulation. Obes Rev. 2011 Jan;12(1):14-25. doi: 10.1111/j.1467-789X.2010.00716.x. PMID 20122134
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Parolin ML, Chesley A, Matsos MP, Spriet LL, Jones NL, Heigenhauser GJ. Regulation of skeletal muscle glycogen phosphorylase and PDH during maximal intermittent exercise. Am J Physiol. 1999 Nov;277(5):E890-900. doi: 10.1152/ajpendo.1999.277.5.E890. PMID 10567017
- [Background] Jensen J, Jebens E, Brennesvik EO, Ruzzin J, Soos MA, Engebretsen EM, O'Rahilly S, Whitehead JP. Muscle glycogen inharmoniously regulates glycogen synthase activity, glucose uptake, and proximal insulin signaling. Am J Physiol Endocrinol Metab. 2006 Jan;290(1):E154-E162. doi: 10.1152/ajpendo.00330.2005. Epub 2005 Aug 23. PMID 16118249
- [Background] Derave W, Hansen BF, Lund S, Kristiansen S, Richter EA. Muscle glycogen content affects insulin-stimulated glucose transport and protein kinase B activity. Am J Physiol Endocrinol Metab. 2000 Nov;279(5):E947-55. doi: 10.1152/ajpendo.2000.279.5.E947. PMID 11052948
- [Background] Casey A, Constantin-Teodosiu D, Howell S, Hultman E, Greenhaff PL. Metabolic response of type I and II muscle fibers during repeated bouts of maximal exercise in humans. Am J Physiol. 1996 Jul;271(1 Pt 1):E38-43. doi: 10.1152/ajpendo.1996.271.1.E38. PMID 8760079
- [Background] Holloszy JO. Exercise-induced increase in muscle insulin sensitivity. J Appl Physiol (1985). 2005 Jul;99(1):338-43. doi: 10.1152/japplphysiol.00123.2005. PMID 16036907
- [Background] Devlin JT, Hirshman M, Horton ED, Horton ES. Enhanced peripheral and splanchnic insulin sensitivity in NIDDM men after single bout of exercise. Diabetes. 1987 Apr;36(4):434-9. doi: 10.2337/diab.36.4.434. PMID 3102297
- [Background] Gibala MJ, Little JP. Physiological basis of brief vigorous exercise to improve health. J Physiol. 2020 Jan;598(1):61-69. doi: 10.1113/JP276849. Epub 2019 Dec 20. PMID 31691289
- [Background] Cochran AJ, Percival ME, Tricarico S, Little JP, Cermak N, Gillen JB, Tarnopolsky MA, Gibala MJ. Intermittent and continuous high-intensity exercise training induce similar acute but different chronic muscle adaptations. Exp Physiol. 2014 May 1;99(5):782-91. doi: 10.1113/expphysiol.2013.077453. Epub 2014 Feb 14. PMID 24532598
- [Background] Bogdanis GC, Nevill ME, Lakomy HK, Boobis LH. Power output and muscle metabolism during and following recovery from 10 and 20 s of maximal sprint exercise in humans. Acta Physiol Scand. 1998 Jul;163(3):261-72. doi: 10.1046/j.1365-201x.1998.00378.x. PMID 9715738
- [Background] Sabag A, Little JP, Johnson NA. Low-volume high-intensity interval training for cardiometabolic health. J Physiol. 2022 Mar;600(5):1013-1026. doi: 10.1113/JP281210. Epub 2021 Apr 18. PMID 33760255
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- [Background] Dey KC, Zakrzewski-Fruer JK, Smith LR, Jones RL, Bailey DP. Interrupting sitting acutely attenuates cardiometabolic risk markers in South Asian adults living with overweight and obesity. Eur J Appl Physiol. 2024 Apr;124(4):1163-1174. doi: 10.1007/s00421-023-05345-7. Epub 2023 Nov 11. PMID 37950762
- [Background] Larsen RN, Kingwell BA, Sethi P, Cerin E, Owen N, Dunstan DW. Breaking up prolonged sitting reduces resting blood pressure in overweight/obese adults. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):976-82. doi: 10.1016/j.numecd.2014.04.011. Epub 2014 May 2. PMID 24875670
- [Background] Wongpipit W, Zhang X, Miyashita M, Wong SH. Interrupting Prolonged Sitting Reduces Postprandial Glucose Concentration in Young Men With Central Obesity. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e791-e802. doi: 10.1210/clinem/dgaa834. PMID 33186451
- [Background] Peddie MC, Bone JL, Rehrer NJ, Skeaff CM, Gray AR, Perry TL. Breaking prolonged sitting reduces postprandial glycemia in healthy, normal-weight adults: a randomized crossover trial. Am J Clin Nutr. 2013 Aug;98(2):358-66. doi: 10.3945/ajcn.112.051763. Epub 2013 Jun 26. PMID 23803893
- [Background] Benatti FB, Ried-Larsen M. The Effects of Breaking up Prolonged Sitting Time: A Review of Experimental Studies. Med Sci Sports Exerc. 2015 Oct;47(10):2053-61. doi: 10.1249/MSS.0000000000000654. PMID 26378942
- [Background] Loh R, Stamatakis E, Folkerts D, Allgrove JE, Moir HJ. Effects of Interrupting Prolonged Sitting with Physical Activity Breaks on Blood Glucose, Insulin and Triacylglycerol Measures: A Systematic Review and Meta-analysis. Sports Med. 2020 Feb;50(2):295-330. doi: 10.1007/s40279-019-01183-w. PMID 31552570
- [Background] Cavalot F, Petrelli A, Traversa M, Bonomo K, Fiora E, Conti M, Anfossi G, Costa G, Trovati M. Postprandial blood glucose is a stronger predictor of cardiovascular events than fasting blood glucose in type 2 diabetes mellitus, particularly in women: lessons from the San Luigi Gonzaga Diabetes Study. J Clin Endocrinol Metab. 2006 Mar;91(3):813-9. doi: 10.1210/jc.2005-1005. Epub 2005 Dec 13. PMID 16352690
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Pappas C, Kandaraki EA, Tsirona S, Kountouras D, Kassi G, Diamanti-Kandarakis E. Postprandial dysmetabolism: Too early or too late? Hormones (Athens). 2016 Jul;15(3):321-344. doi: 10.14310/horm.2002.1697. PMID 27838603
- [Background] O'Keefe JH, Bell DS. Postprandial hyperglycemia/hyperlipidemia (postprandial dysmetabolism) is a cardiovascular risk factor. Am J Cardiol. 2007 Sep 1;100(5):899-904. doi: 10.1016/j.amjcard.2007.03.107. Epub 2007 Jun 26. PMID 17719342
- [Background] Trost SG, Owen N, Bauman AE, Sallis JF, Brown W. Correlates of adults' participation in physical activity: review and update. Med Sci Sports Exerc. 2002 Dec;34(12):1996-2001. doi: 10.1097/00005768-200212000-00020. PMID 12471307
- [Background] Akins JD, Crawford CK, Burton HM, Wolfe AS, Vardarli E, Coyle EF. Inactivity induces resistance to the metabolic benefits following acute exercise. J Appl Physiol (1985). 2019 Apr 1;126(4):1088-1094. doi: 10.1152/japplphysiol.00968.2018. Epub 2019 Feb 14. PMID 30763169
- [Background] Ekelund U, Steene-Johannessen J, Brown WJ, Fagerland MW, Owen N, Powell KE, Bauman A, Lee IM; Lancet Physical Activity Series 2 Executive Committe; Lancet Sedentary Behaviour Working Group. Does physical activity attenuate, or even eliminate, the detrimental association of sitting time with mortality? A harmonised meta-analysis of data from more than 1 million men and women. Lancet. 2016 Sep 24;388(10051):1302-10. doi: 10.1016/S0140-6736(16)30370-1. Epub 2016 Jul 28. PMID 27475271
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] DiPietro L, Al-Ansari SS, Biddle SJH, Borodulin K, Bull FC, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Willumsen JF. Advancing the global physical activity agenda: recommendations for future research by the 2020 WHO physical activity and sedentary behavior guidelines development group. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):143. doi: 10.1186/s12966-020-01042-2. PMID 33239105
- [Background] King WC, Chen JY, Courcoulas AP, Mitchell JE, Wolfe BM, Patterson EJ, Inabnet WB, Dakin GF, Flum DR, Cook B, Belle SH. Objectively-measured sedentary time and cardiometabolic health in adults with severe obesity. Prev Med. 2016 Mar;84:12-8. doi: 10.1016/j.ypmed.2015.12.007. Epub 2015 Dec 24. PMID 26724517
- [Background] Honda T, Chen S, Yonemoto K, Kishimoto H, Chen T, Narazaki K, Haeuchi Y, Kumagai S. Sedentary bout durations and metabolic syndrome among working adults: a prospective cohort study. BMC Public Health. 2016 Aug 26;16(1):888. doi: 10.1186/s12889-016-3570-3. PMID 27562190
- [Background] Dempsey PC, Biddle SJH, Buman MP, Chastin S, Ekelund U, Friedenreich CM, Katzmarzyk PT, Leitzmann MF, Stamatakis E, van der Ploeg HP, Willumsen J, Bull F. New global guidelines on sedentary behaviour and health for adults: broadening the behavioural targets. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):151. doi: 10.1186/s12966-020-01044-0. PMID 33239026
- [Background] Pinto AJ, Bergouignan A, Dempsey PC, Roschel H, Owen N, Gualano B, Dunstan DW. Physiology of sedentary behavior. Physiol Rev. 2023 Oct 1;103(4):2561-2622. doi: 10.1152/physrev.00022.2022. Epub 2023 Jun 16. PMID 37326297
- [Background] Wanner M, Richard A, Martin B, Faeh D, Rohrmann S. Associations between self-reported and objectively measured physical activity, sedentary behavior and overweight/obesity in NHANES 2003-2006. Int J Obes (Lond). 2017 Jan;41(1):186-193. doi: 10.1038/ijo.2016.168. Epub 2016 Sep 28. PMID 27677618
- [Background] Prince SA, Elliott CG, Scott K, Visintini S, Reed JL. Device-measured physical activity, sedentary behaviour and cardiometabolic health and fitness across occupational groups: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2019 Apr 2;16(1):30. doi: 10.1186/s12966-019-0790-9. PMID 30940176
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680